CLINICAL TRIAL: NCT00719940
Title: Randomized Controlled Clinical Trial of Efficacy and Safety of Individual Cognitive Behavioral Therapy (CBT) Within the Setting of the Structured Therapy Program sTCP (Structured Tinnitus Care Program) in Patients With Tinnitus Aurium
Brief Title: Tinnitus Treatment by Structured Cognitive Behavioral Therapy
Acronym: TCP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Zenner, H.P., M.D., Professor & Chairman, Dept. ORL, University of Tuebingen, Germany, University Hospital, University of Tuebingen, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCP00/04; BMBF 01EZ0506: Dekonet;; Mediceon: Benchmarking project
Record Dates: First submitted 2008-06-16; First posted 2008-07-22 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2008-06

CONDITIONS: Tinnitus
Keywords: tinnitus, cognitive behavioral therapy, CBT
MeSH Terms: conditions — Tinnitus; Color Vision Defects | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cognitive behavioral therapy
  Interventions: Behavioral: Cognitive behavioral therapy
- 2 (Placebo Comparator): Waiting group
  Interventions: Other: Waiting group

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — 1-15 individual sessions of 50-60 min. to apply 1-15 manualized tinnitus specific cognitive behavioral therapy interventions structured by the tinnitus care disease management program
  Other Names: tinnitus care program
  Arms: 1
Other: Waiting group — No intervention
  Other Names: tinnitus care program
  Arms: 2

SUMMARY:
Test of hypothesis that in contrast to non-treatment tinnitus specific cognitive behavioral therapy intervention procedures that are manualized and structured within the disease management program TCP are effective.

DETAILED DESCRIPTION:
Intervention:

Individual application of structured and tinnitus specific cognitive behavioral therapy intervention procedures in the clinical setting of the structured therapy program "tinnitus care program (TCP)"

Duration of intervention per patient: 1-15 treatment sessions plus self treatment up to 16 weeks

Control intervention: Waiting group (16 weeks)

ELIGIBILITY:
Key Inclusion Criteria:

* Persistent and stable tinnitus of more than 11 weeks
* Gap between audiometric tinnitus matching and subjective tinnitus loudness rating scale

Key Exclusion Criteria:

* Psychiatric or neurological comorbidity
* Tinnitus as concomitant symptom of an otherwise treatable disease
* Drug treatment for tinnitus 24 hrs. prior or during therapy

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2000-10; Primary Completion 2004-10 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Validated tinnitus questionaire (TF Goebel and Hiller 1992); validated tinnitus change rating scale (TC, Zenner and de Maddalena 2005) | Last session

SECONDARY OUTCOMES:
Tinnitus loudness (TL), validated 6-point numeric verbal rating scale; tinnitus annoyance (TA), validated 8-point numeric verbal rating scale | last therapy session

CONTACTS AND LOCATIONS:
Overall Officials: Hans P. Zenner, M.D., Principal Investigator — Universität Tübingen
Locations (4):
- Germany (4):
  - Tinnitus Care Center, Aschaffenburg
  - Tinnitus Care Center, Frankfurt
  - Dept. ORL, University of Tuebingen, Tübingen
  - Private Practice, Tübingen

REFERENCES:
- [Result] Zenner HP, De Maddalena H. Validity and reliability study of three tinnitus self-assessment scales: loudness, annoyance and change. Acta Otolaryngol. 2005 Nov;125(11):1184-8. doi: 10.1080/00016480510012282. PMID 16353397
- [Derived] Zenner HP, Vonthein R, Zenner B, Leuchtweis R, Plontke SK, Torka W, Pogge S, Birbaumer N. Standardized tinnitus-specific individual cognitive-behavioral therapy: a controlled outcome study with 286 tinnitus patients. Hear Res. 2013 Apr;298:117-25. doi: 10.1016/j.heares.2012.11.013. Epub 2012 Dec 31. PMID 23287811